CLINICAL TRIAL: NCT02528045
Title: Efficacy of Surgical Treatment of Vitrectomy and Scleral Shortening for Macular Hole Retinal Detachment or Myopic Traction Maculopathy
Brief Title: Vitrectomy and Scleral Shortening for Macular Hole Retinal Detachment or Myopic Traction Maculopathy
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Kyorin Eye Center, Kyorin University
Other Study IDs: Kyorineye017
Record Dates: First submitted 2015-08-16; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Macular Hole Retinal Detachment; Myopic Traction Maculopathy
Keywords: Myopic traction maculopathy
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Vitrectomy with scleral shortening

SUMMARY:
The medical records of 16 eyes of 16 patients with macular hole retinal detachment or myopic traction maculopathy who received viterctomy including internal limiting membrane peeling and scleral shorting surgery were reviewed. Best-corrected visual acuity, axial length, retinal reattachment and macular hole closure, the shape of staphyloma determined by optical coherence tomography and 3-dimensional magnetic resonance imaging were assessed.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were patients who had highly myopic eyes with macular hole retinal detachment to myopic traction maculopathy

Exclusion Criteria:

* The patients with follow-up less than 6 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent vitrectomy with scleral shortening for macular hole retinal detachment or myopic traction maculopathy
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Visual acuity before and after surgery | 6 months
  Comparison with logarithm of Minimum Angle of Resolution (logMAR) vision

SECONDARY OUTCOMES:
Retinal reattachment | 6 months
  Retinal reattachment or resolution of myopic traction maculopathy

CONTACTS AND LOCATIONS:
Overall Officials: Akito Hirakata, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Makoto Inoue, Mitaka, Tokyo, Japan